CLINICAL TRIAL: NCT01968824
Title: Efficacy of Brachial Plexus Block in Post-Operative Pain Control After Distal Upper Extremity Fracture: A Prospective Randomized Study
Brief Title: Brachial Plexus Block in Post-Op Pain Control After Distal Upper Extremity Fracture: A Prospective Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S12-02386
Record Dates: First submitted 2013-10-14; First posted 2013-10-24 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Pain
Keywords: pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General Anesthesia (No Intervention): general anesthesia only
- Brachial Plexus Nerve Block (Experimental): brachial plexus nerve block
  Interventions: Procedure: Brachial Plexus Nerve Block

INTERVENTIONS:
Procedure: Brachial Plexus Nerve Block — The brachial plexus will be visualized under ultrasound and a 22 gauge, 3.5 inch needle will be used. 20 cc of bupivicaine will be injected around the brachial plexus after confirming negative aspiration every 5 cc
  Arms: Brachial Plexus Nerve Block

SUMMARY:
Despite the plethora of literature suggesting that regional blockade provides adequate andimproved postoperative pain control, function and improved intraoperative and postoperative safety in proximal upper extremity surgery, little is known of its benefits for the treatment of forearm and distal radius fractures . The purpose of this randomized, prospective, study is to determine if brachial plexus blockade with general anesthesia is superior to general anesthesia alone in immediate and long-term pain control in patients undergoing operative fixation of distal upper extremity fractures.

DETAILED DESCRIPTION:
The purpose of this study is to compare two (2) different types of anesthesia treatments that are used during surgery for broken arms for post-surgery pain relief. One group will receive general anesthesia (state of total unconsciousness) the other group will get sedation (medicine injected into patient's vein that helps patient fall asleep), and a nerve block (injection of anesthetic drug into the nerves going to patient's arm in order to make patient's arm numb).

Both forms of anesthesia are used for a variety of surgeries to the arm including shoulder and elbow surgeries. Currently it is thought that there are advantages and disadvantages to both types. The advantage of not using the nerve block in addition to general anesthesia (current standard or care) is that it decreases the potential risk for bleeding, infection and nerve injury. Alternatively, the advantage of using the nerve block with sedation (research-related procedure) is that it can potentially offer better post-operative pain control. This study will examine whether there is added benefit with the addition of nerve block for anesthesia for decreasing pain after surgical treatment of lower arm fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years old.
2. Male or Female
3. All racial and ethnic groups
4. Fractures and fracture/dislocations of the elbow, forearm, wrist and hand
5. Montaggia and Galleazzi variants
6. Patients who opt for surgical treatment of their fractures.
7. Patients who consent to be randomized.
8. Patients who are willing to follow-up for a minimum of 52 weeks.

Exclusion Criteria:

1. Patients younger than 18 years old.
2. Patients who are unwilling to follow-up for a minimum of 52 weeks.
3. Limitation in upper extremity function that would affect outcome scoring
4. Neurologic condition that could interfere with pain sensation
5. Patients with a contraindication to one of the anesthesia protocols
6. Patients who refuse a specific anesthesia protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Post-Operative Pain | 2 weeks
  post-operative pain will be measured at various time points

CONTACTS AND LOCATIONS:
Overall Officials: Nirmal C Tejwani, MD, Principal Investigator — NYU Hospital for Joint Diseases
Locations (1):
- New York University Langone Medical Center, New York, New York, United States